CLINICAL TRIAL: NCT01286467
Title: A PHASE 1 STUDY TO EVALUATE THE SAFETY, PHARMACOKINETICS, AND PHARMACODYNAMICS OF PF 04449913, AN ORAL HEDGEHOG INHIBITOR, ADMINISTERED AS SINGLE AGENT IN SELECT SOLID TUMORS
Brief Title: A Study Of PF-04449913 Administered Alone In Select Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: B1371002
Record Dates: First submitted 2011-01-14; First posted 2011-01-31 (Estimated); Results first posted 2024-03-06 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2023-08

CONDITIONS: Solid Tumors
Keywords: PF-04449913; Hedgehog Inhibitor; Solid tumor; Pharmacokinetics; Safety; Pharmacodynamics
MeSH Terms: interventions — glasdegib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: PF-04449913

INTERVENTIONS:
Drug: PF-04449913 — Escalating dose of PF-04449913 administered as tablets PO QD in 28-day cycles

SUMMARY:
This study examines the effect of a small molecule inhibitor to the Sonic Hedgehog pathway on select solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological diagnosis of advanced/metastatic solid tumor
* Adequate Bone Marrow Function
* Adequate Renal Function
* Adequate Liver Function

Exclusion Criteria:

* Patients with known symptomatic brain metastases requiring steroids
* Current active treatment on another clinical trial
* Major surgery or radiation therapy within 4-weeks of starting study treatment

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2011-05-11 (Actual); Primary Completion 2012-05-10 (Actual); Study Completion 2012-12-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (9):
- United States (9):
  - Keck Hospital of University of Southern California, Los Angeles, California
  - Los Angeles County-University of Southern California Medical Center, Los Angeles, California
  - University of Southern California/Norris Comprehensive Cancer Center/Investigational Drug Service, Los Angeles, California
  - University of Southern California/Norris Comprehensive Cancer Center, Los Angeles, California
  - Anschutz Cancer Pavilion, Aurora, Colorado
  - University of Colorado Denver, Aurora, Colorado
  - University of Colorado Hospital, Aurora, Colorado
  - Brigham and Women's Hospital (BWH), Boston, Massachusetts
  - Dana-Farber Cancer Institute (DFCI), Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Fostvedt LK, Shaik N, Martinelli G, Wagner AJ, Ruiz-Garcia A. Exposure-response modeling of the effect of glasdegib on cardiac repolarization in patients with cancer. Expert Rev Clin Pharmacol. 2021 Jul;14(7):927-935. doi: 10.1080/17512433.2021.1925538. Epub 2021 May 18. PMID 33993815
- [Derived] Wagner AJ, Messersmith WA, Shaik MN, Li S, Zheng X, McLachlan KR, Cesari R, Courtney R, Levin WJ, El-Khoueiry AB. A phase I study of PF-04449913, an oral hedgehog inhibitor, in patients with advanced solid tumors. Clin Cancer Res. 2015 Mar 1;21(5):1044-51. doi: 10.1158/1078-0432.CCR-14-1116. Epub 2014 Nov 11. PMID 25388167
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1371002&StudyName=A%20Study%20Of%20PF-04449913%20Administered%20Alone%20In%20Select%20Solid%20Tumors

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All enrolled participants were assigned to PF-04449913 dose escalation cohorts.
Groups:
- PF-04449913 80 mg: Participants received oral single agent PF-04449913 tablets 80 milligram (mg) once daily for 25 days in Cycle 1 followed by 3 days without treatment for the purpose of pharmacokinetic (PK) assessments, and for 28 days in Cycles 2 and beyond, i.e. up to a maximum of 14 treatment cycles (one treatment cycle was defined as 28 days).
- PF-04449913 160 mg: Participants received oral single agent PF-04449913 tablets 160 mg once daily for 25 days in Cycle 1 followed by 3 days without treatment for the purpose of PK assessments, and 28 days in Cycles 2 and beyond, i.e. up to a maximum of 14 treatment cycles (one treatment cycle was defined as 28 days).
- PF-04449913 320 mg: Participants received oral single agent PF-04449913 tablets 320 mg once daily for 25 days in Cycle 1 followed by 3 days without treatment for the purpose of PK assessments, and 28 days in Cycles 2 and beyond i.e. up to a maximum of 14 treatment cycles (one treatment cycle was defined as 28 days).
- PF-04449913 640 mg: Participants received oral single agent PF-04449913 tablets 640 mg once daily for 25 days in Cycle 1 followed by 3 days without treatment for the purpose of PK assessments, and 28 days in Cycles 2 and beyond, i.e. up to a maximum of 14 treatment cycles (one treatment cycle was defined as 28 days).
Period: Overall Study
Arm/Group | PF-04449913 80 mg | PF-04449913 160 mg | PF-04449913 320 mg | PF-04449913 640 mg
Started | 4 | 4 | 7 | 8
Completed | 0 | 0 | 0 | 0
Not Completed | 4 | 4 | 7 | 8
Not completed — Death | 1 | 1 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 1
Not completed — Disease progression | 3 | 2 | 2 | 3
Not completed — Adverse Event | 0 | 1 | 2 | 3
Not completed — Study drug stop longer than 14 days | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants
Groups:
- Total: Total of all reporting groups
Arm/Group | PF-04449913 80 mg | PF-04449913 160 mg | PF-04449913 320 mg | PF-04449913 640 mg | Total
Number analyzed (Participants) | 4 | 4 | 7 | 8 | 23
Age, Customized [Count of Participants; unit: Participants]
  18 to 44 years | 2 | 1 | 0 | 0 | 3
  45 to 64 years | 2 | 1 | 4 | 5 | 12
  Greater than or equal to (>=) 65 years | 0 | 2 | 3 | 3 | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 1 | 2 | 2 | 9
  Male | 0 | 3 | 5 | 6 | 14

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With First Cycle Dose Limiting Toxicities (DLTs)
Description: Any DLT event in Cycle 1: (1) Grade 4 neutropenia lasting more than 7 days; (2) Febrile neutropenia; (3) Grade >=3 neutropenic infection; (4) Grade >=3 thrombocytopenia with bleeding; (5) Grade 4 thrombocytopenia lasting more than 7 days; (6) Grade >=3 non-hematologic toxicity; (7) Failure to deliver at least 80% of the planned doses due to toxicities attributable to PF-04449913
Time Frame: Baseline up to end of Cycle 1 (Study Day 28)
Population: Per-Protocol Analysis Set: all enrolled participants who received at least 1 dose of study medication and did not have major treatment deviations during Cycle 1.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-04449913 80 mg | PF-04449913 160 mg | PF-04449913 320 mg | PF-04449913 640 mg
Number analyzed (Participants) | 4 | 3 | 6 | 6
Participants | 0 | 0 | 0 | 2

2. Secondary Outcome: Percentage of Participants With Treatment-emergent Adverse Events (AEs), by National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) (Version 4.0) Grade
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Treatment-emergent AEs are events occurred between first dose of study drug and up to 28 days after last dose that were absent before treatment or that worsened relative to pretreatment state. If the same participant in a given treatment had more than one occurrence in the same preferred term event category, only the worst CTCAE grade was reported. Grades as per NCI CTCAE, v4.0 were classified as: Grade 1- mild, Grade 2- moderate, Grade 3- severe, Grade 4- life threatening, and Grade 5- death.
Time Frame: Baseline up to 28 days post last dose of study medication (maximum duration: 14 cycles [each cycle of 28 days])
Population: Safety Analysis Set: all enrolled participants who received at least 1 dose of study medication.
Measure: Number; unit: percentage of participants
Arm/Group | PF-04449913 80 mg | PF-04449913 160 mg | PF-04449913 320 mg | PF-04449913 640 mg
Number analyzed (Participants) | 4 | 4 | 7 | 8
percentage of participants
  Any AEs, Grade 1 | 0.0 | 0.0 | 14.3 | 0.0
  Any AEs, Grade 2 | 50.0 | 50.0 | 42.9 | 12.5
  Any AEs, Grade 3 | 25.0 | 25.0 | 14.3 | 87.5
  Any AEs, Grade 4 | 0.0 | 0.0 | 14.3 | 0.0
  Any AEs, Grade 5 | 25.0 | 25.0 | 14.3 | 0.0
  Any AEs, Total | 100.0 | 100.0 | 100.0 | 100.0

3. Secondary Outcome: Percentage of Participants With Treatment-related AEs, by NCI CTCAE (Version 4.0) Grade
Description: An AE was any untoward medical occurrence attributed to study drug in a participant who received study drug. Treatment-related AEs are events that were assessed by the investigator as related to study medication. If the same participant in a given treatment had more than one occurrence in the same preferred term event category, only the worst CTCAE grade was reported. Grades as per NCI CTCAE, v4.0 were classified as: Grade 1- mild, Grade 2- moderate, Grade 3- severe, Grade 4- life threatening, and Grade 5- death.
Time Frame: Baseline up to 28 days post last dose of study medication (maximum duration: 14 cycles [each cycle of 28 days])
Population: Safety Analysis Set: all enrolled participants who received at least 1 dose of study medication.
Measure: Number; unit: percentage of participants
Arm/Group | PF-04449913 80 mg | PF-04449913 160 mg | PF-04449913 320 mg | PF-04449913 640 mg
Number analyzed (Participants) | 4 | 4 | 7 | 8
percentage of participants
  Any AEs, Grade 1 | 50.0 | 25.0 | 42.9 | 0.0
  Any AEs, Grade 2 | 25.0 | 50.0 | 57.1 | 25.0
  Any AEs, Grade 3 | 0.0 | 0.0 | 0.0 | 62.5
  Any AEs, Grade 4 | 0.0 | 0.0 | 0.0 | 0.0
  Any AEs, Grade 5 | 0.0 | 0.0 | 0.0 | 0.0
  Any AEs, Total | 75.0 | 75.0 | 100.0 | 87.5

4. Secondary Outcome: Hedgehog Biomarker Modulation: Relative GLI1 Gene Expression (Ratio) to Baseline for Normal Skin on Cycle 1/Day 15
Description: Ribonucleic acid (RNA) was extracted from skin samples and complementary deoxyribonucleic acid (cDNA) was prepared. Gene expression was measured using custom Taqman low density array (TLDA) cards run on the Applied Biosystems ViiATM 7 system. The ratio for each participant at each dosing level was calculated at C1D15 to baseline assay readout (C1D1), and the mean of it is reported in this outcome measure.
Time Frame: Baseline and Cycle 1/Day 15
Population: Pharmacodynamic (PD) Analysis Set: all enrolled participants who received at least 1 dose of study medication, and had baseline and at least 1 on-treatment PD result.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | PF-04449913 80 mg | PF-04449913 160 mg | PF-04449913 320 mg | PF-04449913 640 mg
Number analyzed (Participants) | 3 | 3 | 4 | 5
ratio | 0.1 (0.01) | 0.1 (0.09) | 0.1 (0.04) | 0.1 (0.06)

5. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) on Cycle 1/Day 1
Description: Cmax of PF-04449913 on Cycle 1/Day 1 has been reported.
Time Frame: Pre dose, 1, 2, 4, 6, 10 and 24 hours post dose on Cycle 1/Day 1
Population: PK Analysis Set: all treated participants who had at least 1 of the PK parameters of interest. N=number of participants evaluable for the outcome measure
Measure: Mean (Standard Deviation); unit: nanogram/milliliter (ng/mL)
Arm/Group | PF-04449913 80 mg | PF-04449913 160 mg | PF-04449913 320 mg | PF-04449913 640 mg
Number analyzed (Participants) | 4 | 4 | 7 | 8
nanogram/milliliter (ng/mL) | 1161 (389) | 1126 (949) | 2624 (611) | 6299 (2661)

6. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) on Cycle 1/Day 25
Description: Cmax of PF-04449913 on Cycle 1/Day 25 has been reported.
Time Frame: Pre dose, 1, 2, 4, 10, 24, 48, 72 and 96 hours post dose on Cycle 1/Day 25
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | PF-04449913 80 mg | PF-04449913 160 mg | PF-04449913 320 mg | PF-04449913 640 mg
Number analyzed (Participants) | 4 | 3 | 6 | 4
ng/mL | 1373 (542) | 1567 (475) | 3363 (1716) | 4913 (992)

7. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) on Cycle 1/Day 1
Description: Tmax of PF-04449913 on Cycle 1/Day 1 has been reported.
Time Frame: Pre dose, 1, 2, 4, 6, 10 and 24 hours post dose on Cycle 1/Day 1
Population: as for outcome 5
Measure: Median (Full Range); unit: hours
Arm/Group | PF-04449913 80 mg | PF-04449913 160 mg | PF-04449913 320 mg | PF-04449913 640 mg
Number analyzed (Participants) | 4 | 4 | 7 | 8
hours | 1.5 [1 to 2.2] | 2 [1 to 8] | 2.1 [1 to 4] | 2 [1 to 4]

8. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) on Cycle 1/Day 25
Description: Tmax of PF-04449913 on Cycle 1/Day 25 has been reported.
Time Frame: Pre dose, 1, 2, 4, 10, 24, 48, 72 and 96 hours post dose on Cycle 1/Day 25
Population: as for outcome 5
Measure: Median (Full Range); unit: hours
Arm/Group | PF-04449913 80 mg | PF-04449913 160 mg | PF-04449913 320 mg | PF-04449913 640 mg
Number analyzed (Participants) | 4 | 3 | 6 | 4
hours | 1 [0.9 to 2] | 2 [2 to 10] | 2 [1 to 10] | 4 [1 to 10]

9. Secondary Outcome: Area Under the Curve From Time Zero to End of Dosing Interval (AUCtau) on Cycle 1/Day 1
Description: AUCtau of PF-04449913 on Cycle 1/Day 1 has been reported. AUCtau is defined as area under the curve from time 0 to tau, where tau is the dosing interval of 24 hours.
Time Frame: Pre dose, 1, 2, 4, 6, 10 and 24 hours post dose on Cycle 1/Day 1
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: nanogram*hour/milliliter (ng*hr/mL)
Arm/Group | PF-04449913 80 mg | PF-04449913 160 mg | PF-04449913 320 mg | PF-04449913 640 mg
Number analyzed (Participants) | 4 | 4 | 7 | 8
nanogram*hour/milliliter (ng*hr/mL) | 10510 (3948) | 12540 (8583) | 31160 (11140) | 62550 (18031)

10. Secondary Outcome: Area Under the Curve From Time Zero to End of Dosing Interval (AUCtau) on Cycle 1/Day 25
Description: AUCtau of PF-04449913 on Cycle 1/Day 25 has been reported. AUCtau is defined as area under the curve from time 0 to tau, where tau is the dosing interval of 24 hours.
Time Frame: Pre dose, 1, 2, 4, 10, 24, 48, 72 and 96 hours post dose on Cycle 1/Day 25
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | PF-04449913 80 mg | PF-04449913 160 mg | PF-04449913 320 mg | PF-04449913 640 mg
Number analyzed (Participants) | 4 | 3 | 6 | 4
ng*hr/mL | 13930 (6967) | 18670 (5050) | 46670 (20336) | 70600 (19636)

11. Secondary Outcome: Plasma Decay Half-life (t1/2) on Cycle 1/Day 25
Description: Plasma decay half-life is the time measured for the plasma concentration to decrease by one half.
Time Frame: Pre dose, 1, 2, 4, 10, 24, 48, 72 and 96 hours post dose on Cycle 1/Day 25
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | PF-04449913 80 mg | PF-04449913 160 mg | PF-04449913 320 mg | PF-04449913 640 mg
Number analyzed (Participants) | 4 | 3 | 6 | 4
hours | 19 (5) | 21 (6.7) | 21 (4.9) | 18 (4.3)

12. Secondary Outcome: Apparent Oral Clearance (CL/F) on Cycle 1/Day 25
Description: Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes.
Time Frame: Pre dose, 1, 2, 4, 10, 24, 48, 72 and 96 hours post dose on Cycle 1/Day 25
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: liter/hour (L/hr)
Arm/Group | PF-04449913 80 mg | PF-04449913 160 mg | PF-04449913 320 mg | PF-04449913 640 mg
Number analyzed (Participants) | 4 | 3 | 6 | 4
liter/hour (L/hr) | 7.2 (4.2) | 9.1 (2.9) | 8.0 (3.5) | 9.6 (2.5)

13. Secondary Outcome: Apparent Volume of Distribution (Vz/F) on Cycle 1/Day 25
Description: Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug.
Time Frame: Pre dose, 1, 2, 4, 10, 24, 48, 72 and 96 hours post dose on Cycle 1/Day 25
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: liter (L)
Arm/Group | PF-04449913 80 mg | PF-04449913 160 mg | PF-04449913 320 mg | PF-04449913 640 mg
Number analyzed (Participants) | 4 | 3 | 6 | 4
liter (L) | 182 (69) | 286 (146) | 234 (93) | 249 (88)

14. Secondary Outcome: Accumulation Ratio (Rac) on Cycle 1/Day 25
Description: Accumulation ratio was calculated as AUCtau at steady state (Cycle 1/Day 25)/AUCtau on Study Day 1
Time Frame: Pre dose, 1, 2, 4, 6, 10 and 24 hours post dose on Cycle 1/Day 1, and pre dose, 1, 2, 4, 10, 24, 48, 72 and 96 hours post dose on Cycle 1/Day 25
Population: as for outcome 5
Measure: Median (Full Range); unit: ratio
Arm/Group | PF-04449913 80 mg | PF-04449913 160 mg | PF-04449913 320 mg | PF-04449913 640 mg
Number analyzed (Participants) | 4 | 3 | 6 | 4
ratio | 1.4 [0.9 to 1.6] | 2.2 [1.3 to 4.4] | 1.7 [0.6 to 2.9] | 1.6 [0.7 to 1.8]

15. Secondary Outcome: Average Concentration at Steady State (Cavg) on Cycle 1/Day 25
Time Frame: Pre dose, 1, 2, 4, 10, 24, 48, 72 and 96 hours post dose on Cycle 1/Day 25
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | PF-04449913 80 mg | PF-04449913 160 mg | PF-04449913 320 mg | PF-04449913 640 mg
Number analyzed (Participants) | 4 | 3 | 6 | 4
ng/mL | 580 (290) | 777 (211) | 1942 (848) | 2943 (820)

16. Secondary Outcome: Number of Participants With Increase From Baseline in Corrected QT Using Fridericia's Formula (QTcF) Interval
Description: Triplicate 12-lead electrocardiogram (ECG) measurements (each recording separated by approximately 2 minutes) were performed and average was calculated. The time from electrocardiogram Q wave to the end of the T wave corresponding to electrical systole (QT) was corrected for heart rate (QTc). QTc using Fridericia's formula (QTcF) was calculated. Participants with maximum increase from baseline of less than (<) 30 millisecond (msec), 30 to <60 msec and >=60 msec were summarized.
Time Frame: Baseline up to Cycle 14 (each cycle 28 days)
Population: QTc Analysis Set: all enrolled participants who had at least 1 ECG assessment after receiving at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | PF-04449913 80 mg | PF-04449913 160 mg | PF-04449913 320 mg | PF-04449913 640 mg
Number analyzed (Participants) | 4 | 4 | 7 | 8
participants
  QTcF, maximum increase from baseline: <30 msec | 3 | 4 | 4 | 2
  QTcF, maximum increase from baseline: 30-<60 msec | 1 | 0 | 2 | 5
  QTcF, maximum increase from baseline: >=60 msec | 0 | 0 | 1 | 1

17. Secondary Outcome: Number of Participants With Decrease From Baseline in QTcF Interval
Description: Triplicate 12-lead ECG measurements (each recording separated by approximately 2 minutes) were performed and average was calculated. QTcF was calculated. Participants with maximum decrease from baseline of <30 msec, 30 to <60 msec and >=60 msec were summarized.
Time Frame: Baseline up to Cycle 14 (each cycle 28 days)
Population: as for outcome 16
Measure: Number; unit: participants
Arm/Group | PF-04449913 80 mg | PF-04449913 160 mg | PF-04449913 320 mg | PF-04449913 640 mg
Number analyzed (Participants) | 4 | 4 | 7 | 8
participants
  QTcF, maximum decrease from baseline: <30 msec | 4 | 4 | 6 | 4
  QTcF, maximum decrease from baseline: 30-<60 msec | 0 | 0 | 0 | 0
  QTcF, maximum decrease from baseline: >=60 msec | 0 | 0 | 0 | 0

18. Secondary Outcome: Number of Participants With Post-baseline QTcF Interval Greater Than or Equal to 500 Msec
Description: Triplicate 12-lead ECG measurements (each recording separated by approximately 2 minutes) were performed and average was calculated. Participants with post-baseline absolute QTcF values >=500 msec were summarized.
Time Frame: Baseline up to Cycle 14 (each cycle 28 days)
Population: as for outcome 16
Measure: Number; unit: participants
Arm/Group | PF-04449913 80 mg | PF-04449913 160 mg | PF-04449913 320 mg | PF-04449913 640 mg
Number analyzed (Participants) | 4 | 4 | 7 | 8
participants | 0 | 0 | 1 | 0

19. Secondary Outcome: Percentage of Participants With Objective Response
Description: Percentage of participants with objective response based on assessment of confirmed complete response (CR) or confirmed partial response (PR) according to Response Evaluation Criteria in Solid Tumors (RECIST) 1.1. Confirmed responses were those that persisted on repeat imaging study at least 4 weeks after initial documentation of response. CR was defined as complete disappearance of all target lesions with the exception of nodal disease. PR was defined as >=30% decrease under baseline of the sum of diameters of all target measurable lesions.
Time Frame: Baseline up to Cycle 14 (each cycle 28 days)
Population: Efficacy Analysis Set: all enrolled participants who received at least 1 dose of study medication.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | PF-04449913 80 mg | PF-04449913 160 mg | PF-04449913 320 mg | PF-04449913 640 mg
Number analyzed (Participants) | 4 | 4 | 7 | 8
percentage of participants | 0 [0.0 to 60.2] | 0 [0.0 to 60.2] | 0 [0.0 to 41.0] | 0 [0.0 to 36.9]

20. Secondary Outcome: Progression-Free Survival (PFS)
Description: Time from Cycle 1/Day 1 to first documentation of disease progression or to death due to any cause, whichever occurred first. Progression was defined using RECIST 1.1 as 20% increase in the sum of diameters of target measurable lesions above the smallest sum observed, with a minimum absolute increase of 5 mm. PFS (days) was calculated as (first event date minus the date of first dose of study medication plus 1).
Time Frame: Baseline up to Cycle 14 (each cycle 28 days)
Population: This OM was planned for expansion cohort only. Since none of the participants were enrolled in expansion cohort, no data was collected for progression free survival and thus the outcome measure was not performed.
Arm/Group | PF-04449913 80 mg | PF-04449913 160 mg | PF-04449913 320 mg | PF-04449913 640 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0

21. Secondary Outcome: Time to Progression (TTP)
Description: Time from Cycle 1/Day 1 to first documentation of disease progression. Progression was defined using RECIST 1.1 as 20% increase in the sum of diameters of target measurable lesions above the smallest sum observed, with a minimum absolute increase of 5 mm. TTP (days) was calculated as (first event date minus the date of first dose of study medication plus 1).
Time Frame: Baseline up to Cycle 14 (each cycle 28 days)
Population: This OM was planned for expansion cohort only. Since none of the participants were enrolled in expansion cohort, no data was collected for time to progression and thus the outcome measure was not performed.
Arm/Group | PF-04449913 80 mg | PF-04449913 160 mg | PF-04449913 320 mg | PF-04449913 640 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0

22. Secondary Outcome: Duration of Response (DR)
Description: Duration from date of first documentation of objective response to date of first documentation of disease progression or death. Progression was defined using RECIST 1.1 as 20% increase in the sum of diameters of target measurable lesions above the smallest sum observed, with a minimum absolute increase of 5 mm. DR was calculated as (the date of the first documentation of objective tumor progression or death due to cancer minus the date of the first objective response that was subsequently confirmed plus 1).
Time Frame: Baseline up to Cycle 14 (each cycle 28 days)
Population: This OM was planned for expansion cohort only. Since none of the participants were enrolled in expansion cohort, no data was collected for duration of response and thus the outcome measure was not performed.
Arm/Group | PF-04449913 80 mg | PF-04449913 160 mg | PF-04449913 320 mg | PF-04449913 640 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a serious AE (SAE). However, what are presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | PF-04449913 80 mg | PF-04449913 160 mg | PF-04449913 320 mg | PF-04449913 640 mg
Serious Adverse Events (participants affected / at risk) | 2/4 | 2/4 | 3/7 | 3/8
Other Adverse Events (participants affected / at risk) | 4/4 | 4/4 | 7/7 | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PF-04449913 80 mg (N=4) | PF-04449913 160 mg (N=4) | PF-04449913 320 mg (N=7) | PF-04449913 640 mg (N=8)
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Chills (General disorders) | 0 | 0 | 1 | 0
Disease progression (General disorders) | 0 | 1 | 1 | 0
Pain (General disorders) | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 1 | 0
Peritonitis bacterial (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 1 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PF-04449913 80 mg (N=4) | PF-04449913 160 mg (N=4) | PF-04449913 320 mg (N=7) | PF-04449913 640 mg (N=8)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1
Leukopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 1 | 0 | 2
Sinus tachycardia (Cardiac disorders) | 1 | 0 | 1 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Eye pain (Eye disorders) | 1 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 2
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1 | 2
Abdominal rigidity (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Ascites (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 5
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 4 | 5
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Lip dry (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 1 | 3 | 4
Parotid gland inflammation (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 3 | 2
Asthenia (General disorders) | 0 | 0 | 0 | 1
Chest pain (General disorders) | 0 | 0 | 1 | 0
Chills (General disorders) | 0 | 1 | 0 | 1
Fatigue (General disorders) | 2 | 1 | 4 | 6
Malaise (General disorders) | 0 | 0 | 0 | 1
Mucosal inflammation (General disorders) | 0 | 0 | 0 | 1
Oedema peripheral (General disorders) | 0 | 1 | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 2 | 0 | 0
Respiratory tract infection viral (Infections and infestations) | 0 | 0 | 0 | 1
Sinusitis (Infections and infestations) | 1 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 2 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 1 | 0 | 1
Blood bilirubin increased (Investigations) | 1 | 0 | 2 | 2
Blood creatinine increased (Investigations) | 0 | 0 | 1 | 2
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 0 | 1
Blood uric acid increased (Investigations) | 0 | 0 | 0 | 1
Electrocardiogram QT interval abnormal (Investigations) | 0 | 0 | 1 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 0 | 1
Neutrophil count decreased (Investigations) | 1 | 0 | 0 | 0
Weight decreased (Investigations) | 0 | 1 | 1 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1 | 3 | 5
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 2 | 4
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Muscle atrophy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1 | 2
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 3 | 5
Dysgeusia (Nervous system disorders) | 3 | 2 | 6 | 4
Headache (Nervous system disorders) | 1 | 0 | 0 | 1
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 0 | 0
Memory impairment (Nervous system disorders) | 0 | 1 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 1 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 0 | 1 | 0
Depression (Psychiatric disorders) | 1 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 1 | 1 | 1
Mental status changes (Psychiatric disorders) | 0 | 0 | 0 | 1
Proteinuria (Renal and urinary disorders) | 0 | 0 | 1 | 1
Menstruation irregular (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Prostatitis (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 3
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 0 | 2
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.